CLINICAL TRIAL: NCT01062906
Title: The Effect of Intravenous Lidocaine on Short-term Outcomes After Laparoscopic Cholecystectomy
Brief Title: Intravenous Lidocaine for Laparoscopic Cholecystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Francesco Carli, McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GEN#08-021
Record Dates: First submitted 2010-02-03; First posted 2010-02-04 (Estimated); Last update posted 2011-01-13 (Estimated); Status verified 2010-02

CONDITIONS: Postoperative Pain; Opioid Consumption
Keywords: intravenous lidocaine; postoperative pain; laparoscopic surgery; opioids; opioids side-effects
MeSH Terms: conditions — Pain, Postoperative | interventions — Lidocaine; Fentanyl

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (Placebo Comparator): The control group receives intravenous fentanyl at the induction of anesthesia followed by a continuous infusion of lidocaine during the surgery.
  Interventions: Drug: Fentanyl
- Lidocaine (Active Comparator): The Lidocaine group will receive lidocaine as bolus at the induction of anesthesia followed by a continuous infusion of lidocaine until the end of surgery
  Interventions: Drug: Lidocaine

INTERVENTIONS:
Drug: Lidocaine — 1.5 mg/Kg as bolus and a continuous infusion of 2mg/Kg/hr until the end of surgery (closure of the skin)
  Arms: Lidocaine
Drug: Fentanyl — Fentanyl 3 mcg/Kg as bolus at the induction and a continuous infusion of normal saline (NaCl 0.9%) until the end of surgery (skin closure)
  Arms: Control

SUMMARY:
Intravenous lidocaine has been shown to have analgesic, antinflammatory, antihyperalgesic, antithrombotics and neuroprotective properties. In a previous study conducted in patients undergoing laparoscopic cholecystectomy under general anesthesia with desflurane and fentanyl, intraoperative i.v. infusion of lidocaine spared opioids consumption in the recovery room by 30%.

The purpose of this study was to determine if an i.v. infusion of lidocaine without intraoperative opioids would reduce the amount of fentanyl to the same extent and opioids-related side effects.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing laparoscopic cholecystectomy

Exclusion Criteria:

* age <18 yr or > 85 yr,
* ASA physical status 3 and greater, history of hepatic failure (Child & Pug A-C),
* renal failure (creatinine outside the normal range) or cardiac failure (NYHA I-IV),
* Adams-Stoke syndrome,
* severe degrees of sinoatrial, atrioventricular or intraventricular block,
* organ transplant,
* diabetes mellitus type 1 and 2,
* morbid obesity (BMI > 40),
* chronic use of opioids and beta-blockers,
* known seizures,
* severe mental impairment,
* allergy to local anesthetics and to all the medications used in the study, or
* inability to understand pain assessment.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2010-03; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Fentanyl consumption (measured as fentanyl equivalents -mcg) | postoperative day 0 (day of surgery before beeing discharged home) and 24 hr after the end of surgery

SECONDARY OUTCOMES:
Pain, Static and Dynamic | On postoperative day 0 (day of surgey before beeing discharged home) and 24 hrs after the end of surgery
Opioids side-effects | On postoperative day 0 (before beeing discharged home) and at 24 hrs after the end of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Franco Carli, MD, professor, Principal Investigator — McGill University Healt Centre, Department of Anesthesia
Locations (1):
- McGill University Health Centre, Montreal General Hospital, Montreal, Quebec, Canada

REFERENCES:
- [Background] Lauwick S, Kim DJ, Michelagnoli G, Mistraletti G, Feldman L, Fried G, Carli F. Intraoperative infusion of lidocaine reduces postoperative fentanyl requirements in patients undergoing laparoscopic cholecystectomy. Can J Anaesth. 2008 Nov;55(11):754-60. doi: 10.1007/BF03016348. PMID 19138915